CLINICAL TRIAL: NCT01587352
Title: A Phase 2 Study of Vorinostat (NSC 701852) in Metastatic Uveal Melanoma
Brief Title: Vorinostat in Treating Patients With Metastatic Melanoma of the Eye
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Institut Curie Paris (Unknown); Memorial Sloan Kettering Cancer Center (Other); Moffitt Cancer Center P2C (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-00860; NCI-2012-00860 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 12-027; CUMC-IRBAAAO5917; AAAO5917; MSKCC-12-027; 9111 (Other: Memorial Sloan Kettering Cancer Center); 9111 (Other: CTEP); N01CM00100 (NIH); N01CM62206 (NIH); P30CA008748 (NIH); U01CA069856 (NIH); UM1CA186689 (NIH)
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Uveal Melanoma; Stage IV Uveal Melanoma AJCC v7
MeSH Terms: conditions — Uveal Melanoma | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (vorinostat) (Experimental): Patients receive vorinostat PO BID for 3 days weekly for 4 weeks. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Vorinostat

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Vorinostat — Given PO
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase II trial studies how well vorinostat works in treating patients with melanoma of the eye that has spread to other parts of the body (metastatic). Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the overall objective response rate (RR) to vorinostat in patients with metastatic uveal melanoma.

SECONDARY OBJECTIVES:

I. Overall survival (OS). II. Progression free survival (PFS). III. To determine the tolerability of vorinostat in patients with metastatic uveal melanoma.

EXPLORATORY OBJECTIVES:

I. To correlate clinical outcome with changes in histone acetylation status by immunohistochemistry.

II. To correlate clinical outcome with changes in known proliferation and apoptotic markers including Ki67 by immunohistochemistry and BIM, survivin, c-myc, Mcl-1, cleaved PARP, gamma-H2AX and RAD51 by western blot.

III. To assess for changes in pathways such as the MAPK pathway with treatment. IV. To describe the evolution of circulating cell-free, tumor-derived deoxyribonucleic acid (DNA) levels measured by pyrophosphorolysis activated polymerization (PAP) in plasma of patients under treatment for metastatic uveal melanoma.

V. To correlate overall objective RR with GNAQ, GNA11, SF3B1 and BAP1 mutational status.

OUTLINE:

Patients receive vorinostat orally (PO) twice daily (BID) for 3 days weekly for 4 weeks. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic histologically or cytologically confirmed uveal melanoma. (If histologic or cytologic confirmation of the primary is not available, confirmation of the primary diagnosis of uveal melanoma by the treating investigator can be clinically obtained, as per standard practice for uveal melanoma). Pathologic confirmation of diagnosis will be performed at Columbia University, Memorial Sloan-Kettering Cancer Center (MSKCC) or Vanderbilt University Medical Center
* Patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Age >= 18 years. Because limited dosing or adverse event data are currently available on the use of vorinostat in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric single-agent trials, if applicable
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9.0 g/dL not requiring transfusions within the past 2 weeks
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN); =< 3 x institutional ULN if the patient has Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN if no liver metastasis present; =< 5 x institutional ULN if liver metastases are present
* Creatinine =< 1.5 mg/dL
* Ability to understand and the willingness to sign a written informed consent document
* Vorinostat is toxic to the developing human fetus. For this reason and because Class D agents are known to be teratogenic, women of child-bearing potential and men must agree to use effective contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of vorinostat administration

Exclusion Criteria:

* Patients may have had any number of prior therapies. At least 3 weeks must have elapsed since the last dose of systemic therapy. At least 6 weeks must have elapsed if the last regimen included BCNU or mitomycin C. At least 6 weeks must have elapsed if the last regimen included an anti-CTLA4 antibody. Patients must have experienced disease progression on their prior therapy in the opinion of the treating investigator
* Patients who are receiving any other investigational agents
* Patients with active or untreated brain metastases. Treated brain metastases must have been stable for at least 2 months
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat
* Patients receiving HDAC inhibitors or compounds with HDAC inhibitor like activity, such as valproic acid, are ineligible. Patients who have received such agents may enroll on this study after a 14-day washout period
* Patients on warfarin will be excluded from the trial if they cannot be switched to an acceptable alternative medication (i.e. low molecular weight heparin [LMWH]). Prolongation of prothrombin time (PT) and International Normalized Ratio (INR) were observed in patients receiving vorinostat concomitantly with coumarin-derivative anticoagulants
* Pregnant women are excluded from this study because vorinostat is a Class D agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with vorinostat, breastfeeding should be discontinued if the mother is treated with vorinostat
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy will be eligible unless the CD4 count is < 200 cells/mm^3 within one month of study enrollment (as requested by Cancer Therapy Evaluation Program [CTEP]). These patients are at increased risk of lethal infections when treated with marrow-suppressive therapy
* A second malignancy requiring active therapy
* No concomitant anti-cancer chemotherapy or other systemic drugs. Palliative radiation therapy will be allowed as long as the patient meets all other eligibility criteria
* Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption
* Corrected QT interval (QTc) > 475 milliseconds
* Patients who cannot swallow capsules

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-05-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate in patients with uveal melanoma | Up to 3 years
  Defined as the rate of complete and partial responses. The response rate along with 90% confidence interval will be estimated.

SECONDARY OUTCOMES:
Overall survival | From start of treatment to death or last follow-up will be estimated, assessed up to 3 years
  Overall survival curves will be generated using Kaplan-Meier methodology.
Progression free survival | From start of treatment to date of progression, death or last follow-up will be estimated, assessed up to 3 years
  Progression-free survival curves will be generated using Kaplan-Meier methodology.
Incidence of toxicities | Up to 3 years
  Assessed by National Cancer Institute Common Toxicity Criteria 4.0. Toxicity will be reported by type, frequency and severity.

OTHER OUTCOMES:
Gnaq mutation status | Up to day 15
  Associations of each unique mutation status with overall response will be assessed using Fisher's exact test.
GNA11 mutation status | Up to day 15
  Associations of each unique mutation status with overall response will be assessed using Fisher's exact test.
BAP1 mutation status | Up to day 15
  Associations of each unique mutation status with overall response will be assessed using Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander N Shoushtari, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee